CLINICAL TRIAL: NCT03371394
Title: Body Composition Monitoring in Valvular Heart Disease: Association With Clinical Status and Impact on Prognosis
Brief Title: Fluid Status in Valvular Heart Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Dr. Andreas Kammerlander, MD, Medical University of Vienna
Other Study IDs: BCMinVHD-2439
Record Dates: First submitted 2017-12-07; First posted 2017-12-13 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Valvular Heart Disease; Fluid Overload; Cardiovascular Risk Factor
MeSH Terms: conditions — Heart Valve Diseases; Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- median 1
  Interventions: Other: no intervention
- median 2
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
By bioelectrical impedance spectroscopy (BIS) association of fluid status in patients with valvular heart disease and cardiovascular outcome will be assessed.

DETAILED DESCRIPTION:
Volume overload and abnormal fluid distribution are hallmarks in the syndromes of acute and chronic heart failure (HF) as well as valvular heart disease (VHD). Most patients, at some point in their disease progression, present acutely to an emergency department, where they will typically show symptoms of progressive volume overload.

Most patients respond well to standard diuretic therapy, usually at the costs of impaired renal function. Based on the assumption that clinically overt fluid overload is the result of progressive fluid accumulation, current European Society of Cardiology (ESC) and American College of Cardiology Foundation/American Heart Association (ACCF/AHA) guidelines recommend a correction of volume status using diuretics, to reduce the total fluid volume. However there is no consensus on how to define fluid overload quantitavely.

In patients undergoing dialysis, bioelectrical impedance spectroscopy / body composition monitoring (BCM) is a well established tool to assess fluid status, allowing quantitative measurement.

This study aims to

1. Establish a database reflecting the fluid status assessed by BCM of patients presenting with valvular heart disease according to current guidelines
2. Monitor fluid status assessed by BCM during increased diuretic treatment in patients presenting with cardiac decompensation due to valvular heart disease
3. Assess the association between severity of valvular heart disease assessed by echocardiography and/or cardiac magnetic resonance imaging, fluid status assessed by BCM, and clinical as well as laboratory parameters assessed during clinical routine
4. Assess the relationship between fluid status assessed by BCM and cardiovascular outcome

ELIGIBILITY:
Inclusion Criteria:

* Valvular stenosis and/or regurgitation of all severities as defined by current recommendations
* informed consent
* willingness to perform follow up visit

Exclusion Criteria:

* <18 years old
* pregnancy
* unwillingness to paricipate

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients Valvular stenosis and/or regurgitation of all severities assessed by current recommendations are eligible for this study.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-12-15 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular outcome | 3 years
  composition of hospitalization due to heart failure and cardiovascular death

SECONDARY OUTCOMES:
Severity of valvular heart disease | baseline
  BCM and association with valvular severity assessed using integrated approach to current guidelines for valvular heart disease
NT-proBNP | baseline
  BCM and association with NT-proBNP
Clinical status (NYHA functional class) | baseline
  BCM and association with NYHA functional class
Renal impairment | baseline
  BCM and association with renal impariment (eGFR)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No